CLINICAL TRIAL: NCT01237353
Title: Pilot Study Evaluating Gastric Re-acidification Using Betaine Hydrochloride in Healthy Volunteers With Pharmacologically Induced Hypochlorhydria
Brief Title: Study of the Ability of Betaine Hydrochloride to Increase Stomach Acid in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GastricpH-6264
Record Dates: First submitted 2010-11-05; First posted 2010-11-09 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-05

CONDITIONS: Pharmacodynamic
MeSH Terms: interventions — Betaine; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- betaine hydrochloride and rabeprazole (Experimental)
  Interventions: Dietary Supplement: betaine hydrochloride; Drug: Rabeprazole

INTERVENTIONS:
Dietary Supplement: betaine hydrochloride — betaine hydrochloride 1500mg po x 1 on day 5
Drug: Rabeprazole — rabeprazole po daily x 5 days

SUMMARY:
In this study the investigators will test a nutritional supplement called betaine hydrochloride to see if it can temporarily increase the stomach acid in healthy volunteers who have decreased stomach acid because they take a medicine called rabeprazole.

DETAILED DESCRIPTION:
Investigators will evaluate the extent and time course of gastric re-acidification after oral betaine HCl in healthy volunteers with pharmacologically-induced hypochlorhydria. After betaine HCl dose, gastric pH will be continuously monitored for 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult with no active medical problems or significant chronic diseases as determined by the study doctor based on history, physical exam;
* BMI between 18.5 - 35 kg/m2;
* Taking no medications 2 weeks before and during the study enrollment, including drugs of abuse, prescription or OTC medications (except acetaminophen);
* Subjects must be able to maintain adequate birth control during the study independent of hormonal contraceptive use;
* Be able to provide written informed consent and comply with requirements of the study;
* Avoid eating grapefruit and drinking grapefruit juice from 7 days before the first study day until completion of the entire study;
* Abstinence from alcoholic beverages, caffeinated beverages and orange juice from 6pm the night before a study day until completion of that study day;
* Fast from food and beverages at least 8 hours prior to the study day;
* Be able to read, speak and understand English

Exclusion Criteria:

* Subjects with a history of gastrointestinal disease including gastroesophageal reflux disease, gastritis, peptic ulcer disease or dyspepsia.
* Subjects with a fasting gastric pH of > 4 (i.e. hypochlorhydria)
* Subjects with history of dysphagia, achalasia, or difficulty swallowing capsules, tablets or pills.
* Subjects on prescription or chronic over-the counter medications (including hormonal contraceptives);
* Subjects with known allergy to study interventions;
* Subjects who smoke tobacco;
* Subjects with ongoing alcohol or illegal drug use;
* Subjects who are pregnant, lactating or attempting to conceive;
* Subjects unable to maintain adequate birth control during the study;
* Subjects unable to follow protocol instructions or protocol criteria.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Benet, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited to one clinical site in the U.S.
Pre-assignment Details: Hypochlorhydria was induced through the administration of 20mg oral rabeprazole twice daily with food for four days prior to study day
Groups:
- Betaine Hydrochloride and Rabeprazole: betaine hydrochloride : betaine hydrochloride 1500mg po x 1 on day 5
  Rabeprazole : rabeprazole po daily x 5 days
Period: Overall Study
Arm/Group | Betaine Hydrochloride and Rabeprazole
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Betaine Hydrochloride and Rabeprazole
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age Continuous [Mean (Full Range); unit: years] | 39.83 [25 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Gastric pH After Administration of Betaine Hydrochloride (HCl)
Description: Gastric pH levels monitored with a Heidelberg pH capsule (HC) which sends real-time signals to a computer system that visually plots intestinal pH on a minute-by-minute basis. When subject's pH remained above 4.0 for at least 15 minutes, a 1500 mg dose of betaine HCl was given orally with 90 mL of water, and gastric pH was continuously monitored for 2 hours.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Betaine Hydrochloride and Rabeprazole
Number analyzed (Participants) | 6
units on a scale | 4.54 (0.46)

2. Secondary Outcome: Duration of Gastric pH Status
Description: When subject's pH remained above 4.0 for at least 15 minutes, a 1500 mg dose of betaine HCl was given orally with 90 mL of water, and gastric pH was continuously monitored for 2 hours
Time Frame: 2 hours after dose of betaine HCl
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Betaine Hydrochloride and Rabeprazole
Number analyzed (Participants) | 6
minutes
  Mean time to pH <3.0 | 6.3 (4.3)
  Mean minutes of pH < 3.0 | 72.5 (32.9)
  Mean minutes of pH < 4.0 | 76.8 (30.4)

ADVERSE EVENTS:
Time Frame: 2 hours after betaine HCl dose, or by report of subject
Arm/Group | Betaine Hydrochloride and Rabeprazole
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No